CLINICAL TRIAL: NCT01567566
Title: The Effect of Hip Stabilizer Muscle Strengthening on Pain and Disability for Patients With Non-specific Low Back Pain: an Outcome-based Randomized Controlled Trial
Brief Title: An Efficacy Study of Exercise Rehabilitation on Pain and Disability for Patients With Non-specific Low Back Pain
Acronym: LBP-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Running Injury Clinic (Other)
Collaborators: WCB Alberta (Unknown); Alberta Health services (Other)
Responsible Party: Principal Investigator, Karen D. Kendall, PhD Candidate, Running Injury Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIC-WCB-001
Record Dates: First submitted 2012-03-27; First posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Low Back Pain, Mechanical
Keywords: home based daily exercise program; local lumbopelvic stabilizer muscles; hip stabilizer muscles; real time ultrasound imaging
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local lumbopelvic stabilizers (Active Comparator)
  Interventions: Other: exercise rehabilitation program
- Local lumbopelvic plus hip stabilizers (Experimental)
  Interventions: Other: exercise rehabilitation program

INTERVENTIONS:
Other: exercise rehabilitation program — 6 week home based exercise rehabilitation program with 6 weekly supervised sessions using real time ultrasound as biofeedback to augment training in both treatment arms
  Other Names: Core stabilization exercises; Hip stabilization exercises

SUMMARY:
The primary objective of this study is to compare the efficacy of two different exercise programs for the reduction of pain and disability in a specific subgroup of NSLBP patients and aims to investigate the additive effect of hip stabilization exercises. The investigators hypothesize that the combined local (segmental) stabilizer and hip stabilizer program (T2) will be more effective in reducing pain and disability in NSLBP patients compared to the local (segmental) stabilizer program (T1).

DETAILED DESCRIPTION:
The secondary objective of this study is to measure the changes in lumbopelvic and hip mechanics for both treatment groups following completion of the exercise programs. We hypothesize that there will be differences observed between groups following the 6wk rehabilitation programs, and that only the group completing the combined local (segmental) stabilizer and hip stabilizer strengthening program (T2) will demonstrate significant differences in mechanics compared to baseline testing.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Unilateral or bilateral NSLBP symptoms for a minimum of 6 weeks
* Current symptoms rated at least a 5/10 on a scaled from 0-10

Exclusion Criteria:

* Symptoms 'red flags' for underlying pathological conditions such as bowel and/or bladder problems, radicular symptoms, night pain
* Scoliosis
* Neurological impairment, discogenic pathology, vestibular disorder
* Pregnancy or within 1 year of giving birth
* Previous or ongoing complications from lower extremity injury or surgery in the past year
* Previous surgery to the lumbar spine or hip
* Use of any radiological interventions or injections such as prolotherapy, corticosteroid, or nerve block in the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity measured by a 10cm visual analogue scale | 6 weeks
  Measures will be taken at baseline, at 3wk follow up, and at 6wk follow up to ivestigate the changes at mid point and following the exercise intervention

SECONDARY OUTCOMES:
Change in biomechanical variables using an eight camera motion capture system | 6 weeks
  Measures will be taken at baseline and at 6wk follow up to ivestigate the changes at mid point and following the exercise intervention
Change in disability score as measured by the Oswestry Disability Questionnaire | 6 weeks
  Measures will be taken at baseline, at 3wk follow up, and at 6wk follow up to ivestigate the changes at mid point and following the exercise intervention

CONTACTS AND LOCATIONS:
Overall Officials: Karen D Kendall, MKin, Principal Investigator — Running Injury Clinic, Faculty of Kinesiology, University of Calgary; Reed Ferber, PhD, Study Director — Running Injury Clinic, Faculty of Kinesiology, University of Calgary
Locations (1):
- Running Injury Clinic, Calgary, Alberta, Canada